CLINICAL TRIAL: NCT02238145
Title: Postmarketing Surveillance Study (as Per § 67 (6) AMG [German Drug Law] of Atrovent® Inhaletten® in Chronic Obstructive Airways Disease
Brief Title: Postmarketing Surveillance Study of Atrovent® Inhaletten® in Chronic Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 244.2492
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Obstructive Airways Disease
  Interventions: Drug: Atrovent® Inhaletten

INTERVENTIONS:
Drug: Atrovent® Inhaletten

SUMMARY:
To obtain further information on the tolerability and efficacy of Atrovent® inhaletten® in the treatment of chronic obstructive airways disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Primarily patients of both gender, older than 30 years,who suffer from chronic obstructive airways disease
* Only patients who had not been treated with Atrovent® within the last year were to be considered for inclusion

Exclusion Criteria:

- Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Atrovent® Inhaletten®

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive airways disease recruited at general practitioners, pneumologists, internists
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 1999-01; Primary Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Investigator assessment of improvement in the clinical picture of the course on a 6-point symptoms profile | Up to 4 weeks after first study drug administration

SECONDARY OUTCOMES:
Investigator assessment of tolerability on a 4-point scale | Up to 4 weeks after first study drug administration
Investigator assessment of efficacy on a 4-point scale | Up to 4 weeks after first study drug administration
Number of patients with adverse drug reactions | Up to 4 weeks after first study drug administration
Number of patients who withdrew from the study | Up to 4 weeks after first study drug administration
Number of patients who changed the concomitant medication | Up to 4 weeks after first study drug administration
Number of patients who continued treatment | Up to 4 weeks after first study drug administration
Patient assessment of tolerability on a 4-point scale | Up to 4 weeks after first study drug administration
Patient assessment of efficacy on a 4-point scale | Up to 4 weeks after first study drug administration